CLINICAL TRIAL: NCT05889962
Title: Effects of Ultrasound-guided Pudendal Nerve Block on Postoperative Pain and Quality of Recovery in Patients Undergoing Hemorrhoidectomy
Brief Title: Ultrasound-guided Pudendal Nerve Block for Pain After Hemorrhoidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N202303039
Record Dates: First submitted 2023-05-02; First posted 2023-06-05 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2023-06

CONDITIONS: Hemorrhoids; Postoperative Pain
MeSH Terms: conditions — Hemorrhoids; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients are randomly allocated into pudendal block group or placebo group. Pudendal block group: Patients will receive pudendal nerve block with ropivacaine.
  Placebo group: Patients will receive pudendal nerve block with normal saline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pudendal block group (Experimental): Receiving bilateral pudendal nerve block with 0.5% ropivacaine (10 ml each side)
  Interventions: Procedure: Pudendal nerve block
- Placebo group (Placebo Comparator): Receiving bilateral pudendal nerve block with normal saline (10 ml each side)
  Interventions: Procedure: Placebo block

INTERVENTIONS:
Procedure: Pudendal nerve block — Patients who are randomized in the pudendal block group will receive bilateral pudendal nerve block with ropivacaine.
  Arms: Pudendal block group
Procedure: Placebo block — Patients who are randomized in the placebo group will receive bilateral pudendal block with normal saline.
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to investigate the effects of ultrasound-guided pudendal nerve block on postoperative pain, opioid consumption, and quality of recovery in patients receiving Ferguson hemorrhoidectomy.

DETAILED DESCRIPTION:
Patients who have symptomatic hemorrhoids undergoing Ferguson hemorrhoidectomy under spinal anesthesia will be randomized to receive bilateral ultrasound-guided pudendal nerve block with 0.5% ropivacaine or normal saline immediately after surgery. In addition, intravenous patient controlled analgesia, NSAIDs, and acetaminophen will be used in all participants for postoperative pain control. Postoperative pain on numerical rating scale (NRS), opioid consumption, quality of recovery (QOR-15), patient's satisfaction, and complications will be recorded at 6, 12, 24, 48 hours and 7 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic hemorrhoids (grade III and grade IV internal hemorrhoids, mixed hemorrhoids, and external hemorrhoids)
* Age 20 to 65 years old
* American Society of Anesthesiologists (ASA) classification I~III
* Receiving Ferguson hemorrhoidectomy under spinal anesthesia

Exclusion Criteria:

* Allergy to local anesthetics or analgesics used in this study
* Drug abuse
* Coagulopathy
* An active infection at the injection site
* Patient refusal
* BMI ≥ 30
* Pregnancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Pain score on the numeric rating scale (NRS) at baseline | Baseline
  NRS ranges from 0 (no pain) to 10 (worst pain)
Postoperative pain score on the numeric rating scale (NRS) at 6 hours | 6 hours after hemorrhoidectomy
  NRS ranges from 0 (no pain) to 10 (worst pain)
Postoperative pain score on the numeric rating scale (NRS) at 12 hours | 12 hours after hemorrhoidectomy
  NRS ranges from 0 (no pain) to 10 (worst pain)
Postoperative pain score on the numeric rating scale (NRS) at 24 hours | 24 hours after hemorrhoidectomy
  NRS ranges from 0 (no pain) to 10 (worst pain)
Postoperative pain score on the numeric rating scale (NRS) at 48 hours | 48 hours after hemorrhoidectomy
  NRS ranges from 0 (no pain) to 10 (worst pain)
Postoperative pain score on the numeric rating scale (NRS) at 7 days | 7 days after hemorrhoidectomy
  NRS ranges from 0 (no pain) to 10 (worst pain)
Opioid consumption at 6 hours | 6 hours after hemorrhoidectomy
  Morphine equivalent dose
Opioid consumption at 12 hours | 12 hours after hemorrhoidectomy
  Morphine equivalent dose
Opioid consumption at 24 hours | 24 hours after hemorrhoidectomy
  Morphine equivalent dose
Opioid consumption at 48 hours | 48 hours after hemorrhoidectomy
  Morphine equivalent dose
Opioid consumption at 7 days | 7 days after hemorrhoidectomy
  Morphine equivalent dose
Quality of recovery at baseline | Baseline
  Quality of recovery-15 questionnaire measures the baseline quality of recovery
Quality of recovery at 24 hours | 24 hours after hemorrhoidectomy
  Quality of recovery-15 questionnaire measures the quality of recovery after surgery
Quality of recovery at 48 hours | 48 hours after hemorrhoidectomy
  Quality of recovery-15 questionnaire measures the quality of recovery after surgery
Quality of recovery at 7 days | 7 days after hemorrhoidectomy
  Quality of recovery-15 questionnaire measures the quality of recovery after surgery

SECONDARY OUTCOMES:
Time to first rescue analgesics | Up to 7 days after hemorrhoidectomy
  Time after hemorrhoidectomy
Time to the first urination | Up to 48 hours after hemorrhoidectomy
  Time after hemorrhoidectomy
Time to the first defecation | Up to 48 hours after hemorrhoidectomy
  Time after hemorrhoidectomy
Patient satisfaction with pain control | 24 hours after hemorrhoidectomy
  0 (worst) to 10 (Best)
Postoperative complications | Up to 7 days after hemorrhoidectomy
  Pudendal nerve block related complications

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Wen Lee, MD, PhD, Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No